CLINICAL TRIAL: NCT07145060
Title: A Randomized Controlled Study of Yiqi Yangyin Formula in the Treatment of Primary Sjogren's Syndrome
Brief Title: A Study of Yiqi Yangyin Formula in the Treatment of Primary Sjogren's Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Luo Jing, Associate chief physician, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-QNQS-07
Record Dates: First submitted 2025-07-04; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Primary Sjögren's Syndrome (pSS)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yiqi Yangyin Formula (Experimental): The herbal prescription for patients eligible for pSS "Qi-Yin deficiency syndrome" , 200 ml twice daily for 12 weeks.
  Interventions: Drug: Yiqi Yangyin Formula
- Yiqi Yangyin Formula placebo (Placebo Comparator): The herbal prescription placebo for patients eligible for pSS "Qi-Yin deficiency syndrome" , 200 ml twice daily for 12 weeks.
  Interventions: Drug: Yiqi Yangyin Formula placebo

INTERVENTIONS:
Drug: Yiqi Yangyin Formula — Yiqi Yangyin Formula,consists of seven Chinese herbal medicines（Table 1）: Rehmanniae Radix (Sheng Di Huang), Lilium brownii (Bai He), Adenophorae Radix (Nan Sha Shen), Fructus Hordei Germinatus (Sheng Mai Ya), Artemisia annua (Qing Hao), Cimicifuga foetida (Sheng Ma) , and Bupleurum chinense(Chai Hu)
  Other Names: The treatment group
  Arms: Yiqi Yangyin Formula
Drug: Yiqi Yangyin Formula placebo — Yiqi Yangyin Formula placebo,has the same appearance, state, and taste as YQYYF, but contains 5% of the ingredients of Yiqi Yangyin Formula
  Other Names: The control group
  Arms: Yiqi Yangyin Formula placebo

SUMMARY:
This project aims to conduct a prospective, randomized, double-blind, controlled clinical study to clarify the efficacy and safety of the YiQi YangYin Formula in treating patients with primary Sjogren's syndrome (pSS) presenting with Qi and Yin deficiency syndrome, with the expectation of providing a scientific basis for the research and development of new traditional Chinese medicine drugs for the effective treatment of pSS.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged18-75 years old (including the critical value), gender not limited;
* Patients meeting the classification criteria of primary Sjogren's syndrome in ACR/EULAR 2016;
* Patients with dry mouth VAS ≥4 and ESSDAI score < 5;
* Patients with positive autoantibodies (ANA or anti-SSA antibodies or anti-SSB antibodies or RF) and/or hyperimmunoglobulinemia or increased erythrocyte sedimentation rate;
* Patients meeting the syndrome of qi and Yin deficiency in traditional Chinese medicine;
* The subjects were informed and voluntarily signed the informed consent form.

Exclusion Criteria:

* Patients with a history of hypersensitivity or intolerance to any investigational therapeutic drug;
* Patients diagnosed with secondary Sjogren's syndrome or combined with other connective tissue diseases;
* Patients with severe lesions in the heart, brain, lungs, liver, kidneys, hematopoietic system, etc., as well as those with malignant tumors or infectious diseases;
* Patients who are pregnant, preparing for pregnancy or breastfeeding;
* Patients who have used cholinergic drugs or artificial tears/saliva in last 1 week;
* Patients who have used hydroxychloroquine, total glycosides of Paeonia lactide, Iguratimod, cyclophosphamide, cyclosporine A, tacrolimus, and azathioprine in last 1 month;
* Patients who have used glucocorticoids, methotrexate or mycophenolate mofetil in last 3 months;
* Patients who have used Leflunomide in last 6 months;
* Patients who have used rituximab in last 6 months, or have used other biological agents (such as tofacitinib) other than rituximab in last 3 months;
* Patients who have participated in or are currently receiving any other experimental drugs or experimental medical devices within the past three months;
* Other situations that researchers consider ineligible for inclusion (such as cognitive impairment, taking psychotropic drugs).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Unstimulated Whole Saliva flow rate (UWS) | week0、week12
  Before the measurement, the participants should avoid eating, drinking, smoking, brushing teeth. and sit still for 10 minutes to collect all the saliva that flows out within 15 minutes in a clean container. The volume will be measured and the salivary secretion rate per unit time will be calculated, which is the UWS (ml/min). UWS ≤ 0.1 ml/min is defined as low UWS.

SECONDARY OUTCOMES:
bilateral Schirmer's test | week0、week12
  Without surface anesthesia, in a quiet and dim environment, bend the standard Schirmer filter paper at the scale and gently place it on the edge of the lower temporal eyelid of the subject. Instruct the subject to gently close their eyes and keep the filter paper for 5 minutes. After 5 minutes, remove the filter paper and measure the wet length. Schirmer≤5 mm/5 min indicates the presence of dry eye syndrome.
EULAR Sjögren Syndrome Patient Reported Index (ESSPRI) | week0、week4、week8、week12
  The ESSRPI is a patient-reported index for Sjogren's syndrome, which includes scores for sjogren's symptoms, limb pain, and physical fatigue. The weights of the three aspects are the same, and each aspect's score ranges from 0 to 10. ESSPRI is defined as the average of these three aspects, with a score range of 0 to 10. The higher the value, the more severe the condition. A symptom state of less than 5 is acceptable to the patient, while a symptom state of ≥5 is unsatisfactory to the patient.
EULAR Sjögren syndrome disease activity index (ESSDAI) | week0、week12
  Low activity is defined as ESSDAI < 5 points, moderate activity as 5≤ESSDAI≤13 points, and high activity as ESSDAI≥14 points
Sjögren's Tool for Assessing Response (STAR) | week12
  It includes the assessment of ESSDAI system involvement, the subjective perception assessment of ESSPRI patients, the functional changes of salivary glands and lacrimal glands, and the evaluation of serological indicators for treatment response. A total score of ≥5 is considered a treatment response.
Composite of Relevant Endpoints for Sjogren Syndrome (CRESS) | week 12
  It includes an assessment of five aspects，at least three out of the five have responded is defined as a response.
erythrocyte sedimentation rate (ESR), C-reactive protein (CRP) | 0week、12week
  conventional inflammatory marks
36-Item Short Form Survey (SF-36) | week0、week12
  The higher the score, the better the quality of life
serum immunoglobulin（IgA、IgM、IgG） | week0、week12
  Compare the differences in the values of various serological indicators between the two groups of patients at the time of enrollment and 12 weeks after treatment, as well as the proportion of improvement and aggravation of serological indicators.
Complement (C3, C4） | week0、week12
  Compare the differences in the values of various serological indicators between the two groups of patients at the time of enrollment and 12 weeks after treatment, as well as the proportion of improvement and aggravation of serological indicators.

CONTACTS AND LOCATIONS:
Overall Officials: Tao Qingwen Tao, Study Chair — China-Japan Friendship Hospital
Locations (1):
- China-Japan friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seror R, Ravaud P, Mariette X, Bootsma H, Theander E, Hansen A, Ramos-Casals M, Dorner T, Bombardieri S, Hachulla E, Brun JG, Kruize AA, Praprotnik S, Tomsic M, Gottenberg JE, Devauchelle V, Devita S, Vollenweider C, Mandl T, Tzioufas A, Carsons S, Saraux A, Sutcliffe N, Vitali C, Bowman SJ; EULAR Sjogren's Task Force. EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI): development of a consensus patient index for primary Sjogren's syndrome. Ann Rheum Dis. 2011 Jun;70(6):968-72. doi: 10.1136/ard.2010.143743. Epub 2011 Feb 22. PMID 21345815
- [Background] Guo N, Wu F, Wu M, Wang Y, Lang Q, Lin X, Feng Y. Progress in the design and quality control of placeboes for clinical trials of traditional Chinese medicine. J Integr Med. 2022 May;20(3):204-212. doi: 10.1016/j.joim.2022.02.005. Epub 2022 Feb 21. PMID 35248517
- [Background] Day SJ, Altman DG. Statistics notes: blinding in clinical trials and other studies. BMJ. 2000 Aug 19-26;321(7259):504. doi: 10.1136/bmj.321.7259.504. No abstract available. PMID 10948038
- [Background] Brito-Zeron P, Theander E, Baldini C, Seror R, Retamozo S, Quartuccio L, Bootsma H, Bowman SJ, Dorner T, Gottenberg JE, Mariette X, Bombardieri S, de Vita S, Mandl T, Ng WF, Kruize AA, Tzioufas A, Vitali C, Buyon J, Izmirly P, Fox R, Ramos-Casals M; Eular Sjogren Syndrome Task Force. Early diagnosis of primary Sjogren's syndrome: EULAR-SS task force clinical recommendations. Expert Rev Clin Immunol. 2016;12(2):137-56. doi: 10.1586/1744666X.2016.1109449. Epub 2015 Dec 22. PMID 26691952
- [Background] Chan AW, Boutron I, Hopewell S, Moher D, Schulz KF, Collins GS, Tunn R, Aggarwal R, Berkwits M, Berlin JA, Bhandari N, Butcher NJ, Campbell MK, Chidebe RCW, Elbourne DR, Farmer AJ, Fergusson DA, Golub RM, Goodman SN, Hoffmann TC, Ioannidis JPA, Kahan BC, Knowles RL, Lamb SE, Lewis S, Loder E, Offringa M, Ravaud P, Richards DP, Rockhold FW, Schriger DL, Siegfried NL, Staniszewska S, Taylor RS, Thabane L, Torgerson DJ, Vohra S, White IR, Hrobjartsson A. SPIRIT 2025 statement: updated guideline for protocols of randomised trials. BMJ. 2025 Apr 28;389:e081477. doi: 10.1136/bmj-2024-081477. PMID 40294953
- [Background] Mentz RJ, Hernandez AF, Berdan LG, Rorick T, O'Brien EC, Ibarra JC, Curtis LH, Peterson ED. Good Clinical Practice Guidance and Pragmatic Clinical Trials: Balancing the Best of Both Worlds. Circulation. 2016 Mar 1;133(9):872-80. doi: 10.1161/CIRCULATIONAHA.115.019902. PMID 26927005
- [Background] Cheng CW, Wu TX, Shang HC, Li YP, Altman DG, Moher D, Bian ZX; CONSORT-CHM Formulas 2017 Group. CONSORT Extension for Chinese Herbal Medicine Formulas 2017: Recommendations, Explanation, and Elaboration. Ann Intern Med. 2017 Jun 27;167(2):112-121. doi: 10.7326/M16-2977. Print 2017 Jul 18. PMID 28654980
- [Background] Fox RI, Fox CM, Gottenberg JE, Dorner T. Treatment of Sjogren's syndrome: current therapy and future directions. Rheumatology (Oxford). 2021 May 14;60(5):2066-2074. doi: 10.1093/rheumatology/kez142. PMID 31034046
- [Background] Bowman SJ, Everett CC, O'Dwyer JL, Emery P, Pitzalis C, Ng WF, Pease CT, Price EJ, Sutcliffe N, Gendi NST, Hall FC, Ruddock SP, Fernandez C, Reynolds C, Hulme CT, Davies KA, Edwards CJ, Lanyon PC, Moots RJ, Roussou E, Giles IP, Sharples LD, Bombardieri M. Randomized Controlled Trial of Rituximab and Cost-Effectiveness Analysis in Treating Fatigue and Oral Dryness in Primary Sjogren's Syndrome. Arthritis Rheumatol. 2017 Jul;69(7):1440-1450. doi: 10.1002/art.40093. Epub 2017 Jun 5. PMID 28296257
- [Background] Ramos-Casals M, Brito-Zeron P, Bombardieri S, Bootsma H, De Vita S, Dorner T, Fisher BA, Gottenberg JE, Hernandez-Molina G, Kocher A, Kostov B, Kruize AA, Mandl T, Ng WF, Retamozo S, Seror R, Shoenfeld Y, Siso-Almirall A, Tzioufas AG, Vitali C, Bowman S, Mariette X; EULAR-Sjogren Syndrome Task Force Group. EULAR recommendations for the management of Sjogren's syndrome with topical and systemic therapies. Ann Rheum Dis. 2020 Jan;79(1):3-18. doi: 10.1136/annrheumdis-2019-216114. Epub 2019 Oct 31. PMID 31672775
- [Background] Brito-Zeron P, Retamozo S, Gheitasi H, Ramos-Casals M. Treating the Underlying Pathophysiology of Primary Sjogren Syndrome: Recent Advances and Future Prospects. Drugs. 2016 Nov;76(17):1601-1623. doi: 10.1007/s40265-016-0659-z. PMID 27844414
- [Background] Brito-Zeron P, Baldini C, Bootsma H, Bowman SJ, Jonsson R, Mariette X, Sivils K, Theander E, Tzioufas A, Ramos-Casals M. Sjogren syndrome. Nat Rev Dis Primers. 2016 Jul 7;2:16047. doi: 10.1038/nrdp.2016.47. PMID 27383445